CLINICAL TRIAL: NCT01853735
Title: Enteral Nutrition in the Open Abdomen
Brief Title: Enteral Feeding in the Post-Injury Open Abdomen
Status: Completed | Type: Observational
Sponsor: Denver Health and Hospital Authority (Other)
Responsible Party: Principal Investigator, Ryan Lawless, Physician, Denver Health and Hospital Authority
Other Study IDs: 13-0077
Record Dates: First submitted 2013-01-15; First posted 2013-05-15 (Estimated); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Trauma to the Abdomen
MeSH Terms: conditions — Abdominal Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- bowel injury, NPO: Patients with bowel injury who remain nil-per-os (fed nothing)
- bowel injury, EN: Patients with bowel injury who are fed by enteral nutrition (EN)
- no bowel injury, NPO: Patients without bowl injury who remain nil-per-os (fed nothing)
- no bowel injury, EN: Patient without bowl injury who are fed by enteral nutrition (EN)

SUMMARY:
The purpose of this study is to determine if Enteral Feeding (EN) in patients with a traumatic bowel injury requiring an open abdomen impacts outcomes. Patients who receive EN will be compared to those who remain nil-per-os (NPO). Additionally, an internal study control will be performed by analyzing concurrent injured patients requiring an open abdomen who did not have a bowel injury.

Specific aims:

Hypothesis 1: EN in patients with a traumatic bowel injury requiring an open abdomen improves fascial closure rate compared to patients who remain NPO.

Hypothesis 2: EN in patients with a traumatic bowel injury requiring an open abdomen reduces infectious complications compared to patients who remain NPO.

Hypothesis 3: EN in patients with a traumatic bowel injury requiring an open abdomen have a lower mortality rate compared to patients who remain NPO.

DETAILED DESCRIPTION:
Fascial closure is determine by the primary physician and should be recorded in the operative record. This record will be accessed to determine if this variable is accomplished. Additionally, any dehiscence complication will be recorded (which would impact the long-term fascial closure rate). Infectious complications (abscess, pneumonia, etc) will be adjudicated by the primary clinician and any record of this in the patient chart will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* All patients with a post-injury open abdomen

Exclusion Criteria:

* Patients to be excluded from analysis include deaths within 24 hours, identification of injury > 24 hours, and those transferred from an outside hospital > 24 hours following initial injury.

Ages: 18 Years to 98 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients requiring an open abdomen following trauma will be prospectively followed.
Sampling Method: Probability Sample
Enrollment: 515 (Actual)
Dates: Start 2013-01; Primary Completion 2022-06-29 (Actual); Study Completion 2022-06-29 (Actual)

PRIMARY OUTCOMES:
fascial closure rate | participants will be followed for their hospital stay, which is on average expected to be 1 month
  physical exam will document fascial closure

SECONDARY OUTCOMES:
mortality | participants will be followed for their hospital stay, which is on average expected to be 1 month
  subject mortality status

OTHER OUTCOMES:
infectious complications | participants will be followed for their hospital stay, which is on average expected to be 1 month
  physical exam and imaging will be reviewed to assess infections

CONTACTS AND LOCATIONS:
Overall Officials: Clay Cothren Burlew, MD, Principal Investigator — Denver Health and Hospital Authority
Locations (1):
- Denver Health Medical Center, Denver, Colorado, United States